CLINICAL TRIAL: NCT03840213
Title: Nutrition and Chemotherapy, Representation and Practice in a Cancer Care Centre (JEUNETCHIMIO)
Brief Title: Nutrition and Chemotherapy
Acronym: JEUNETCHIMIO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institut de Cancérologie de la Loire (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-0101SP; 2019-A00093-54 (Other: ANSM)
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Cancer
Keywords: Chemotherapy; nutrition; self-care; care/caregiver relationship; fasting
MeSH Terms: conditions — Neoplasms; Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing chemotherapy treatment: Patients over 18 years of age, followed at the ICLN day hospital or hospitalized and undergoing chemotherapy treatment
  Interventions: Behavioral: Filling a questionnaire and interviewDescription

INTERVENTIONS:
Behavioral: Filling a questionnaire and interviewDescription — The questionnaire focuses on the dietary practices of patients treated with chemotherapy. It consists of 35 questions, completing an average of 20 minutes.
  Interviews will be conducted with patients who have changed their diet since the beginning of their treatment in order to further develop the results of the quantitative survey.

SUMMARY:
Patients treated for cancer nowadays have many means of information and tend to become more and more involved in their health. The interest of a therapeutic fast with detoxifying or even curative properties, with a specific indication for cancer patients treated by chemotherapy, is nowadays relayed by the media. To date, there are no studies conducted on the scope of this information in cancer patients or on the attitudes of oncologists towards this practice and possible positioning requests from patients.

We hypothesize that the choice of this practice and its modalities are rarely discussed with oncologists, although it may have deleterious repercussions on the patient's health.

We propose a research based on the principles of sociological intervention. Its objectives are a first review of the issue and the establishment of a joint working group, including patients, carers and researchers, which will propose solutions to improve the patient/carer dialogue on this issue.

DETAILED DESCRIPTION:
Patients treated for cancer nowadays have many means of information and tend to become more and more involved in their health. The interest of a therapeutic fast with detoxifying or even curative properties, with a specific indication for cancer patients treated by chemotherapy, is nowadays relayed by the media. To date, there are no studies conducted on the scope of this information in cancer patients or on the attitudes of oncologists towards this practice and possible positioning requests from patients.

We hypothesize that the choice of this practice and its modalities are rarely discussed with oncologists, although it may have deleterious repercussions on the patient's health.

We propose a research based on the principles of sociological intervention. Its objectives are a first review of the issue and the establishment of a joint working group, including patients, carers and researchers, which will propose solutions to improve the patient/carer dialogue on this issue.

ELIGIBILITY:
Inclusion Criteria:

* Major patients, follow-up on Institut de Cancerology Lucien Neuwirth day service chemotherapy treatment
* Patient affiliated or entitled to a social security scheme
* Patient who received informed information about the study
* Patient able to read French

Patients participating in the qualitative study:

Exclusion Criteria:

* Refusal to participate, protected adult person, under guardianship or curatorship
* Person unable to understand the conduct of the study
* Person with a documented history of cognitive or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who intend to practice, or who practice a form of fasting during their chemotherapy treatment will be proposed to participate to a qualitative study to collect more information about their fasting.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-02-20 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients who voluntarily changed their eating habits | 1 year
  Number of patients who voluntarily changed their eating habits will be reported

SECONDARY OUTCOMES:
Number of patients on therapeutic fasting or restrictive diet during chemotherapy treatment | 1 year
  Number of patients on therapeutic fasting or restrictive diet during chemotherapy treatment will be reported
Number of patients using complementary or alternative medicines | 1 year
  Number of patients using complementary or alternative medicines will be reported
Number of patients discussing these different practices with their oncologist | 1 year
  Number of patients discussing these different practices with their oncologist will be reported
Number of patients discussing these different practices with other caregivers | 1 year
  Number of patients discussing these different practices with other caregivers will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fournel, MD, Principal Investigator — Institut de Cancérologie Lucien Neuwirth
Locations (1):
- Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez, France

IPD SHARING:
Plan to Share IPD: No